CLINICAL TRIAL: NCT03635190
Title: Evaluation of the Cardio Flow FreedomFlow™ Orbital Circumferential Atherectomy System to Treat Peripheral Artery Disease
Brief Title: Evaluation of the FreedomFlow™ Orbital Atherectomy System to Treat Peripheral Artery Disease
Acronym: FASTII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardio Flow, Inc. (Industry)
Collaborators: Libra Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010-055
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Results first posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-07

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Diseases; Peripheral Artery Diseases; Arterial Occlusive Diseases; Peripheral Vascular Diseases
MeSH Terms: conditions — Peripheral Arterial Disease; Arterial Occlusive Diseases; Peripheral Vascular Diseases

STUDY DESIGN:
Intervention Model Description: prospective, multi-center, non-randomized single-arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Interventional (Experimental): Orbital Circumferential Atherectomy
  Interventions: Device: Orbital Circumferential Atherectomy

INTERVENTIONS:
Device: Orbital Circumferential Atherectomy — Remove atherosclerotic plaque and modify vessel wall compliance within peripheral arterial vessels. The therapy is intended for patients who are acceptable candidates for percutaneous transluminal atherectomy.
  Other Names: Orbital Atherectomy Atherectomy

SUMMARY:
To evaluate the safety and effectiveness of the Cardio Flow FreedomFlow™ Orbital Circumferential Atherectomy System for atherosclerotic plaque removal and vessel compliance modification in de novo native target lesions in the peripheral vasculature of the lower extremities.

DETAILED DESCRIPTION:
The FAST II study is a prospective, multi-center, non-randomized single-arm trial designed to evaluate the safety and effectiveness of the FreedomFlow™ Orbital Circumferential Atherectomy System in subjects diagnosed with peripheral arterial disease (PAD) of the lower extremities.

The FreedomFlow™ Orbital Circumferential Atherectomy System is a minimally invasive, catheter-based system designed for improving luminal diameter and modifying vessel wall compliance in patients with PAD.

The FreedomFlow™ Orbital Circumferential Atherectomy System is indicated to remove atherosclerotic plaque and modifying vessel wall compliance within peripheral arterial vessels. The therapy is intended for patients who are acceptable candidates for percutaneous transluminal atherectomy.

The objective of the study is to evaluate the safety and effectiveness of the FreedomFlow™ Orbital Circumferential Atherectomy System for atherosclerotic plaque removal and vessel modification in de novo target lesions in the peripheral vasculature of the lower extremities.

ELIGIBILITY:
Subjects must meet all of the following criteria to be eligible for participation in the study:

Inclusion Criteria

1. Age ≥ 18 years old.
2. Subject is a candidate for percutaneous endovascular intervention for peripheral vascular disease in the lower extremity.
3. Objective hemodynamic criteria that subject has a resting ankle-brachial index (ABI) ≤ 0.90 OR a resting toe-brachial index (TBI) of ≤ 0.80 OR ankle pressure of ≤70 mmHg.
4. Clinical presentation of lifestyle limiting claudication, rest pain and/or ischemic wounds as characterized by Rutherford Classification 2, 3, 4, or 5.
5. Disease is located in the common femoral, superficial femoral, popliteal, tibioperoneal, anterior tibial, posterior tibial, and/or peroneal arteries.

   1. De novo target lesion(s) with stenosis ≥70% by visual estimation and/or
   2. Lesion(s) treated by percutaneous transluminal angioplasty (PTA) and/or atherectomy ≥3 months prior with a restenosis ≥70% by visual estimation.
   3. Up to three lesions can be treated at the index procedure provided the cumulative total lesion length is ≤ 20 cm AND all lesions are in the same target leg.
6. Target reference vessel diameter (proximal to and distal to target lesion) is 2 to 8 mm by angiographic visual estimation.
7. At least one patent vessel run-off to the ankle or foot at baseline.
8. The target lesion(s) can be successfully crossed with a commercially available 0.014" atherectomy guidewire without any complications during wiring procedure.
9. Subject signs a written Informed Consent form to participate in the study, prior to any study mandated determinations or procedure.

Subject must be excluded from participation in this study if any of the following criteria are met:

Exclusion Criteria

1. Is female with childbearing potential not taking adequate contraceptives or is currently breastfeeding.
2. Target lesion is within a native graft or synthetic graft.
3. Target lesion is an in-stent restenosis.
4. Target lesion is a chronic total occlusion (CTO) with occlusion length greater than 10 cm and/or with wire crossed sub-intimally. CTO wire placement in true lumen must be confirmed via Intra-vascular ultrasound (IVUS) prior to enrollment.
5. Subject has significant stenosis or occlusion of inflow tract (upstream disease) not successfully treated during the index procedure and prior to treatment of the target lesion.
6. Intra-operative (intra-procedure) clinical or angiographic complication (other than non-flow limiting dissections) attributed to the use of a currently marketed device prior to introduction of the Cardio Flow atherectomy drive shaft.
7. Evidence or history of aneurysmal target vessel.
8. Clinical/angiographic evidence of distal embolization prior to intervention.
9. History of an endovascular procedure or open vascular surgery on the index limb within 30 days prior to the index procedure. Endovascular procedure or open vascular surgery on the non-index limb cannot be staged within 2 weeks prior to the index procedure.
10. Planned endovascular or surgical procedure prior to the subject's 30 day follow up.
11. Signs and symptoms of systemic infection (temperature of ≥ 38.0° Celsius and/or white blood cell count (WBC) of ≥ 12,000 cells/µL) at the time of assessment; Note: If infection is adequately treated and controlled (temperature < 38.0° C and WBC < 12,000 cells/µL) patient may be enrolled.
12. Unstable coronary artery disease or other comorbid condition(s) that, in the judgment of the physician precludes safe percutaneous intervention.
13. Significant acute or chronic kidney disease with a creatinine level > 2.5mg/dL and/or requiring dialysis.
14. Evidence of intracranial or gastrointestinal bleeding, intracranial aneurysm, myocardial infarction or stoke within 2 months of index procedure.
15. Known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated.
16. Subjects in whom anti-platelet, anticoagulant, or thrombolytic therapy is contraindicated.
17. Heparin-induced thrombocytopenia (HIT) not able to use Bivalirudin.
18. Uncorrectable bleeding diathesis, platelet dysfunction, thrombocytopenia with platelet count less than 125,000/mm2, known coagulopathy, or international normalized ratio (INR) > 1.8.
19. Evidence of thrombus within target lesion or thrombolytic therapy within 2 weeks of the index procedure.
20. Has life expectancy < 12 months in the opinion of the investigator.
21. Subject is unwilling or unable to comply with the follow-up study requirements.
22. Subject is currently participating in an investigational drug or another investigational device exemption (IDE) study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fadi Saab, MD, Principal Investigator — Advanced Cardiac & Vascular Amputation Prevention Centers; Thomas P Davis, MD, Principal Investigator — Eastlake Cardiovascular
Locations (13):
- United States (13):
  - Orlando Heart and Vascular Institute, Altamonte Springs, Florida
  - Palm Vascular Center of Broward, LLC, Fort Lauderdale, Florida
  - Cardiovascular Research of North Florida, LLC, Gainesville, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Cardiology Partners Clinical Research Institute, Palm Beach Gardens, Florida
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Cardiovascular Institute of the South, Opelousas, Louisiana
  - Advanced Cardiac & Vascular Centers for Amputation Prevention, Grand Rapids, Michigan
  - Eastlake Cardiovascular, PC, Saint Clair Shores, Michigan
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - Texas Tech University Medical Center, Lubbock, Texas
  - Orion Medical Research, LLC, Pasadena, Texas
  - Cardiovascular Associates of East Texas, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Lesions
Groups:
- Atherectomy Treatment Per Lesion: Measure outcomes of atherectomy treatment based on all lesions treated in 112 patients.
Period: Overall Study
Arm/Group | Atherectomy Treatment Per Lesion
Started | 112; 154 Lesions (Some endpoints were evaluated on a per patient basis and some on a per lesion basis)
Completed | 103; 152 Lesions (2 lesions were not evaluable or results not reported)
Not Completed | 9; 2 Lesions
Not completed — Lost to Follow-up | 4
Not completed — Death | 3
Not completed — Withdrawal by Subject | 1
Not completed — Patient moved and did not return for follow up | 1

BASELINE CHARACTERISTICS:
Population: Some patients had multiple lesions treated. Treatment results for 2 lesions were not evaluable or not reported
Units Other Than Participants: Lesions
Groups:
- Interventional Treatment: 112 patients had 154 lesions treated
Arm/Group | Interventional Treatment
Number analyzed (Participants) | 112
Number analyzed (Lesions) | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Ethnicity not reported for 1 patient
  Participants
    Asian | 1
    Black or African Origin | 16
    Caucasian | 86
    Hispanic or Latino | 7
    Native American or Alaskan Native | 1
    Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 112
Rutherford Classification [Count of Participants; unit: Participants] — Rutherford Classification scale ranges from 1 (normal) to 5 (minor tissue loss). The higher the number the more severe the disease.
  Participants
    2 Moderate Claudication | 9
    3 Severe Claudication | 55
    4 Ischemic Rest Pain | 34
    5 Minor Tissue Loss | 14

OUTCOME MEASURES:

1. Primary Outcome: Technical Success
Description: Defined as the ability of the Cardio Flow FreedomFlow™ Orbital Circumferential Atherectomy System to achieve a residual diameter stenosis ≤50% without adjunctive therapy.
Time Frame: At the time of the index procedure, usually within one hour after starting the procedure
Population: 154 distinct lesions in 112 patients were analyzed
Measure: Count of Units; unit: lesion
Units Other Than Participants: lesion
Groups:
- Site Reported Treatment: Atherectomy treated lesions
  Remove atherosclerotic plaque and modify vessel wall compliance within peripheral arterial vessels.
Arm/Group | Site Reported Treatment
Number analyzed (Participants) | 112
Number analyzed (lesion) | 154
lesion | 144

2. Primary Outcome: Freedom From Major Adverse Events
Description: Primary safety endpoint is freedom from a composite of new onset major adverse events (MAE) at 30-day follow-up as adjudicated by an Independent Clinical Events Committee. This endpoint is evaluated on a per patient basis.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional
Number analyzed (Participants) | 112
Participants | 104

3. Secondary Outcome: Clinical Success
Description: Defined as the ability of the FreedomFlow™ Orbital Circumferential Atherectomy System to achieve a final diameter stenosis <50% immediately post treatment with or without adjunctive therapy, as assessed by an independent Angiographic Core Laboratory.
Time Frame: At index procedure
Measure: Number; unit: lesions
Units Other Than Participants: lesion
Arm/Group | Interventional
Number analyzed (Participants) | 112
Number analyzed (lesion) | 144
lesions | 143

4. Secondary Outcome: Procedure Success
Description: Defined as <50% residual stenosis at target lesion with or without adjunctive therapy, no procedure-related MAE, no device malfunction causing the procedure to be aborted.
Time Frame: At index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional
Number analyzed (Participants) | 112
Participants | 102

5. Secondary Outcome: Ankle Brachia, Index (ABI) Measured at Baseline, 30 Days and 6 Months
Description: ABI measured at baseline, 30 days and 6 months. ABI ranges from 0 to 1, with smaller values indicating more severe disease. Normal ABI is 1.
Time Frame: 30 days and 6 months
Population: Only 107 patients had ABI reported at 30 days and 103 patients had ABI reported at 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interventional
Number analyzed (Participants) | 112
units on a scale
  Baseline ABI | 0.69 (0.22)
  30 day ABI: number analyzed (Participants) | 107
  30 day ABI | 0.90 (0.25)
  6 month ABI: number analyzed (Participants) | 103
  6 month ABI | 0.85 (0.29)

6. Secondary Outcome: Rutherford Classification
Description: Change in Rutherford Classification at 30 days and 6 months. Rutherford scale ranges from 0 to 6 with higher values indicating more severe disease. Rutherford classifications are: 0 Asymptomatic; 1 Mild Claudication; 2 Moderate Claudication; 3 Severe Claudication; 4 Ischemic Rest Pain; 5 Minor Tissue Loss; 6 Major Tissue Loss.
Time Frame: 30 days and 6 months
Population: Only 107 Patients had reported Rutherford Class at 30 days and only 103 Patients had reported Rutherford Class at 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interventional
Number analyzed (Participants) | 112
units on a scale
  Baseline | 3.50 (0.82)
  30 Days: number analyzed (Participants) | 107
  30 Days | 1.00 (1.32)
  6 Months: number analyzed (Participants) | 103
  6 Months | 0.90 (1.29)

7. Secondary Outcome: Vascular Quality of Life Questionnaire (VascuQoL) Administered at Baseline, 30 Days and 6 Months
Description: Patient reported outcomes (PRO, VascuQoL questionnaire) at baseline, 30 days and 6 months. The VascuQoL questionnaire is a validated PRO for lower limb ischemia patients. The range of scores is 1 (worst) to 7 (best)
Time Frame: Baseline, 30 days and 6 months
Population: Only 107 patients had reported VascuQoL at 30 days and only 103 patients had reported VascuQoL at 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interventional
Number analyzed (Participants) | 112
units on a scale
  Baseline VascuQoL | 3.96 (1.42)
  30 day VascuQoL: number analyzed (Participants) | 107
  30 day VascuQoL | 5.33 (1.27)
  6 month VascuQoL: number analyzed (Participants) | 103
  6 month VascuQoL | 5.32 (1.30)

8. Secondary Outcome: Target Lesion and Vessel Revascularization
Description: Clinically driven target lesion revascularization (TLR) at 6 months, target vessel revascularization (TVR) at 30 days and 6 months (as assessed by an independent Angiographic Core Laboratory). Clinically driven target lesion revascularization refers to disease progression that is caused by a recurrence of stenosis at the lesion that was treated; target vessel revascularization refers to disease progression that is caused by a recurrence of stenosis in the same vessel as the treated lesion but at a different site.
Time Frame: 30 days and 6 months
Population: Onlt 103 patients had TLR reported at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional
Number analyzed (Participants) | 112
Participants
  Freedon From TLR at 30 days | 112
  Freedom from TLR at 6 months: number analyzed (Participants) | 109
  Freedom from TLR at 6 months | 103

9. Secondary Outcome: Vessel Patency
Description: Primary patency, primary assisted patency and secondary patency at 30 days and 6 months. Patency will be evaluated on a per lesion basis by duplex ultrasound and evaluated by an independent Vascular Ultrasound Core Laboratory. Restenosis is defined as Peak Systolic Velocity Rate (PSVR) of 2.5. Patency is determined using ultrasound to measure velocity. Patency is indicated for PSVR values < 2.5
Time Frame: 30 days and 6 months
Population: Only 129 lesions had patency reported at 30 days and only 121 lesions had patency reported at 6 months
Measure: Count of Units; unit: lesion
Units Other Than Participants: lesion
Groups:
- Primary Patency; Primary Assisted Patency: Patency will be evaluated by duplex ultrasound and evaluated by an independent Vascular Ultrasound Core Laboratory. The restenosis is defined as PSVR of 2.5.
Arm/Group | Primary Patency | Primary Assisted Patency
Number analyzed (Participants) | 112 | 112
Number analyzed (lesion) | 129 | 129
lesion
  Primary Patency at 30 days | 123 | 128
  Primary Patency at 6 months: number analyzed (lesion) | 121 | 121
  Primary Patency at 6 months | 86 | 113

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Interventional: Atherectomy Treatment
Arm/Group | Interventional
All-Cause Mortality (participants affected / at risk) | 3/112
Serious Adverse Events (participants affected / at risk) | 32/112
Other Adverse Events (participants affected / at risk) | 71/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventional (N=112)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Infection, local (Infections and infestations) | 4 (5)
Target Lesion Revascularization (Vascular disorders) | 4 (4)
Distal Embolization (Vascular disorders) | 3 (3)
Amputation below the knee (Surgical and medical procedures) | 2 (3)
Congestive Heart Failure (Cardiac disorders) | 2 (2)
Infection, systemic (Infections and infestations) | 2 (2)
Non-Target Vessel Revascularization (Vascular disorders) | 2 (2)
Target Vessel Revascularization (Vascular disorders) | 1 (2)
Access Site Hematoma > 6cm (Vascular disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Renal Insufficiency (Renal and urinary disorders) | 1 (1)
Target Vessel Non-target Lesion Revascularization (Vascular disorders) | 1 (1)
Vessel Slow Flow Phenomenon (Vascular disorders) | 1 (1)
Vessel Perforation Type I (Vascular disorders) | 1 (1)
Other (General disorders) | 16 (23)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventional (N=112)
Other (Vascular disorders) | 71 (199) — Non-serious AE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT03635190/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/90/NCT03635190/SAP_001.pdf